CLINICAL TRIAL: NCT01852890
Title: Gemcitabine, Ascorbate, Radiation Therapy for Pancreatic Cancer, Phase I
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Joseph J. Cullen (Other)
Collaborators: Holden Comprehensive Cancer Center (Other); Gateway for Cancer Research (Other)
Responsible Party: Sponsor-Investigator, Joseph J. Cullen, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201310772
Record Dates: First submitted 2013-05-03; First posted 2013-05-14 (Estimated); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Pancreatic Neoplasms
Keywords: Ascorbate; Vitamin C; Radiation; Gemcitabine; Ascorbic Acid
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Ascorbic Acid; Gemcitabine; Radiotherapy; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- 50g Ascorbate (Experimental): This arm is the initial starting dose. The first study participant will be assigned the 50g ascorbate arm.
  * Radiation: Prescribed to either 50 Gy in 25 fractions or at least 50.4 Gy in 28 fractions, based on tumor. Radiation is delivered 1 fraction/day, 5 days a week, for approximately 5 to 6 weeks.
  * Gemcitabine: 600 mg/m2, once weekly for 6 weeks.
  * Ascorbate: 50 grams administered intravenously (by IV) during radiation therapy, for approximately 5 to 6 weeks.
  Interventions: Drug: Ascorbate; Drug: Gemcitabine; Radiation: Radiation therapy
- 75g Ascorbate (Experimental): If the 50g arm is tolerated, the study opens the 75g arm.
  * Radiation: Prescribed to either 50 Gy in 25 fractions or at least 50.4 Gy in 28 fractions, based on tumor. Radiation is delivered 1 fraction/day, 5 days a week, for approximately 5 to 6 weeks.
  * Gemcitabine: 600 mg/m2, once weekly for 6 weeks.
  * Ascorbate: 75 grams administered intravenously (by IV) during radiation therapy, for approximately 5 to 6 weeks.
  Interventions: Drug: Ascorbate; Drug: Gemcitabine; Radiation: Radiation therapy
- 100g Ascorbate (Experimental): If the 75g arm is tolerated, the study opens the 100g arm.
  * Radiation: Prescribed to either 50 Gy in 25 fractions or at least 50.4 Gy in 28 fractions, based on tumor. Radiation is delivered 1 fraction/day, 5 days a week, for approximately 5 to 6 weeks.
  * Gemcitabine: 600 mg/m2, once weekly for 6 weeks.
  * Ascorbate: 100 grams administered intravenously (by IV) during radiation therapy, for approximately 5 to 6 weeks.
  Interventions: Drug: Ascorbate; Drug: Gemcitabine; Radiation: Radiation therapy
- 25g Ascorbate (Experimental): This study arm will only be used if participants cannot tolerate the 50g arm. If participants cannot tolerate 50 grams of Ascorbate, the 25g arm is opened.
  * Radiation: Prescribed to either 50 Gy in 25 fractions or at least 50.4 Gy in 28 fractions, based on tumor. Radiation is delivered 1 fraction/day, 5 days a week, for approximately 5 to 6 weeks.
  * Gemcitabine: 600 mg/m2, once weekly for 6 weeks.
  * Ascorbate: 25 grams administered intravenously (by IV) during radiation therapy, for approximately 5 to 6 weeks.
  Interventions: Drug: Ascorbate; Drug: Gemcitabine; Radiation: Radiation therapy

INTERVENTIONS:
Drug: Ascorbate — Intravenous infusion of high-dose ascorbate
  Other Names: Ascorbic Acid; Vitamin C
Drug: Gemcitabine — Intravenous chemotherapeutic
  Other Names: Gemzar
Radiation: Radiation therapy
  Other Names: External beam radiation therapy; Intensity modulated radiation therapy; IMRT

SUMMARY:
This is a phase 1 (first in man) study testing the safety of adding high dose ascorbate (vitamin C) to standard radiation and chemotherapy for treatment of pancreatic cancer.

DETAILED DESCRIPTION:
This phase 1 study will test the safety of adding high dose ascorbate (vitamin C) to standard chemoradiation. The ascorbate is infused during external beam radiation therapy treatment.

For patients eligible for this trial, standard treatment for their cancer includes radiation therapy combined with weekly gemcitabine (a chemotherapy).

Participants will:

* receive high doses of intravenous (IV) ascorbate during their daily radiation therapy treatments. Radiation treatments are given once a day, Monday through Friday.
* have routine doctor's visits and be asked about any side effects they are experiencing.

This is a phase 1 study that will evaluate the side effects of adding ascorbate to standard therapy. The dose given to a participant will be determined by how well other participants have tolerated ascorbate.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically diagnosed pancreatic adenocarcinoma. Documentation of disease extent by CT scan is required. Radiologically measurable disease is not required.
* Age ≥ 18 years
* ECOG performance status 0, 1, or 2 (Karnofsky > 50%).
* A complete blood count and differential must be obtained within 21 days prior to radiation fraction 1, with adequate bone marrow functions as defined below:

  * Absolute neutrophil count (ANC) ≥ 1500 cells per mm3
  * Platelets ≥ 100,000 per mm3
  * Leukocytes ≥ 3,000 per mm3
* Serum blood chemistries within 21 days of radiation fraction 1, as defined below:

  * Creatinine ≤ 1.5 x UIHC upper limit of normal or creatinine clearance of at least 60 ml/min/1.73 m2 for patients with creatinine levels above institutional normal.
  * Total bilirubin ≤ 2 x UIHC upper limit of normal
  * ALT ≤ 2.5 times the UIHC upper limit of normal
  * AST ≤ 2.5 times the UIHC upper limit of normal
  * PT/INR within normal limits (UIHC)
* Tolerate one test dose (15g) of ascorbate.
* Not pregnant.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* G6PD (glucose-6-phosphate dehydrogenase) deficiency.
* Prior abdominal radiotherapy that would result in overlap of fields. The treating radiation oncologist should review prior RT fields as available.
* Adjuvant therapy (including radiation therapy) within 2 calendar weeks. Toxicities from prior therapy for the malignancy should resolve to grade 1 or less.
* Patients actively receiving insulin are excluded.
* Patients who are on the following drugs and cannot have a drug substitution: flecainide, methadone, amphetamines, quinidine, and chlorpropamide. High dose ascorbate may affect urine acidification and, as a result, may affect clearance rates of these drugs.
* Second malignancy other than non-melanoma skin cancers within the past 5 years.
* Other investigational agents/therapy with the intention to treat the disease under study (observational or imaging trials are acceptable).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, psychiatric illness/social situations, or any other condition that would limit compliance with study requirements as determined by study team members.
* Pregnant or lactating women: The risks of radiation and chemotherapy to a fetus are well documented.
* Known HIV-positive individuals. High-dose ascorbate acid is a known CYP450 3A4 inducer, which results in lower serum levels of antiretroviral drugs. A clinical trial designed to address these interaction issues is more appropriate than this phase 1 study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2019-01-22 (Actual); Study Completion 2025-10-14 (Actual)

PRIMARY OUTCOMES:
Number of grade 3, 4, & 5 adverse events during radiation | Weekly during therapy for up to 10 weeks
  Assess grade 3 and higher adverse events. Evaluate the frequency and severity against the published literature to determine the likely causality between ascorbate and the adverse event(s).

SECONDARY OUTCOMES:
Time to progression | Monthly, up to 10 years post-treatment
  Time from the start of therapy (radiation day 1) to documented disease progression as described by RECIST.
Overall survival | Monthly, up to 10 years post-treatment
  From start of treatment (radiation day 1) until the date of death from any cause.
Number of grade 3, 4, & 5 adverse events post-treatment | every 3 months for 2 years
  Beginning one month after completing radiation therapy, grade 3 and higher adverse events will be assessed. Evaluate the frequency and severity against the published literature to determine the likely causality between ascorbate and the adverse event(s).

CONTACTS AND LOCATIONS:
Overall Officials: Joseph J Cullen, MD, FACS, Principal Investigator — The University of Iowa Hospitals & Clinics
Locations (1):
- The Holden Comprehensive Cancer Center, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared as per approved IRB application and the subject's opt-in preferences. Data will not be provided from subjects who decline data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After completion of primary outcome.
Access Criteria: Interested researchers should contact the study PI. A non-disclosure may need to be filed dependent upon data requested.

REFERENCES:
- [Background] Welsh JL, Wagner BA, van't Erve TJ, Zehr PS, Berg DJ, Halfdanarson TR, Yee NS, Bodeker KL, Du J, Roberts LJ 2nd, Drisko J, Levine M, Buettner GR, Cullen JJ. Pharmacological ascorbate with gemcitabine for the control of metastatic and node-positive pancreatic cancer (PACMAN): results from a phase I clinical trial. Cancer Chemother Pharmacol. 2013 Mar;71(3):765-75. doi: 10.1007/s00280-013-2070-8. Epub 2013 Feb 5. PMID 23381814
- [Background] Du J, Cullen JJ, Buettner GR. Ascorbic acid: chemistry, biology and the treatment of cancer. Biochim Biophys Acta. 2012 Dec;1826(2):443-57. doi: 10.1016/j.bbcan.2012.06.003. Epub 2012 Jun 20. PMID 22728050
- [Background] Cullen JJ. Ascorbate induces autophagy in pancreatic cancer. Autophagy. 2010 Apr;6(3):421-2. doi: 10.4161/auto.6.3.11527. Epub 2010 Apr 15. PMID 20400857
- [Background] Du J, Martin SM, Levine M, Wagner BA, Buettner GR, Wang SH, Taghiyev AF, Du C, Knudson CM, Cullen JJ. Mechanisms of ascorbate-induced cytotoxicity in pancreatic cancer. Clin Cancer Res. 2010 Jan 15;16(2):509-20. doi: 10.1158/1078-0432.CCR-09-1713. Epub 2010 Jan 12. PMID 20068072
- [Result] Mezey E, Potter JJ, French SW, Tamura T, Halsted CH. Effect of chronic ethanol feeding on hepatic collagen in the monkey. Hepatology. 1983 Jan-Feb;3(1):41-4. doi: 10.1002/hep.1840030106. PMID 6295907